CLINICAL TRIAL: NCT04838860
Title: A Phase 2 Study of Intrapatient Siltuximab Dose Escalation in Patients With Idiopathic Multicentric Castleman Disease That Has Progressed After Prior Siltuximab Treatment
Brief Title: Siltuximab In Siltuximab-RElapsed/REfractory Multicentric CAstleman Disease
Acronym: SISREMCAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal Company Decision
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUSA SYL 0002
Record Dates: First submitted 2021-02-25; First posted 2021-04-09 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Multicentric Castleman's Disease
MeSH Terms: conditions — Multi-centric Castleman's Disease | interventions — siltuximab

STUDY DESIGN:
Intervention Model Description: Enrolling in Stage 1a and Stage 1b of this study in parallel will be up to 6 patients each with siltuximab-relapsed or refractory IL-6-driven iMCD and TAFRO-iMCD patients, respectively, who will undergo intrapatient dose escalation of siltuximab beginning with 22 mg/kg q3w, then possibly dose escalating to 33 mg/kg q3w then 44 mg/kg q3w if clinically indicated in the absence of DLT. The justifications for escalating siltuximab doses up to 44 mg/kg q3w will be based on intrapatient dose escalation and DLT assessments as described below.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Parallel Arm of iMCD Patients (Active Comparator): Enrolling in Stage 1a of this study in parallel will be up to 6 patients each with siltuximab-relapsed or refractory IL-6-driven iMCD patients, respectively, who will undergo intrapatient dose escalation of siltuximab beginning with 22 mg/kg q3w, then possibly dose escalating to 33 mg/kg q3w then 44 mg/kg q3w if clinically indicated in the absence of DLT. The justifications for escalating siltuximab doses up to 44 mg/kg q3w will be based on intrapatient dose escalation and DLT assessments as described below.
  Interventions: Drug: Siltuximab
- Parallel Arm of TAFRO-iMCD Patients (Active Comparator): Enrolling in Stage 1b of this study in parallel will be up to 6 patients each with siltuximab-relapsed or refractory IL-6-driven TAFRO-iMCD patients, respectively, who will undergo intrapatient dose escalation of siltuximab beginning with 22 mg/kg q3w, then possibly dose escalating to 33 mg/kg q3w then 44 mg/kg q3w if clinically indicated in the absence of DLT. The justifications for escalating siltuximab doses up to 44 mg/kg q3w will be based on intrapatient dose escalation and DLT assessments as described below.
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — Participants will receive intravenous (IV) infusion of siltuximab 22 mg/kg over 2 hours every 3 weeks, then possibly dose escalating to 33 mg/kg IV over 3 hours +/- 44 mg/kg IV over 4 hours every 3 weeks if clinically indicated in the absence of dose-limiting toxicity.
  Other Names: Sylvant

SUMMARY:
Phase 2 study to investigate the safety, tolerability, and efficacy of administering increased siltuximab doses to patients with iMCD

DETAILED DESCRIPTION:
This is an open-label, two-stage, Phase 2 study to investigate the safety, tolerability, and efficacy of administering increased siltuximab doses to patients with iMCD who progressed with elevated and rising serum C reactive protein (CRP) levels after prior treatment with siltuximab 11 mg/kg every 3 weeks (q3w) without unacceptable toxicity, and is primarily designed to leverage opportunities for intrapatient dose escalation with available clinical, nonclinical, and PK justification as a means to restore or enable disease control.

Enrolling in Stage 1a and Stage 1b of this study in parallel will be up to 6 patients each with siltuximab-relapsed or refractory IL-6-driven iMCD and TAFRO-iMCD patients, respectively, who will undergo intrapatient dose escalation of siltuximab beginning with 22 mg/kg q3w, then possibly dose escalating to 33 mg/kg q3w then 44 mg/kg q3w if clinically indicated in the absence of DLT. The justifications for escalating siltuximab doses up to 44 mg/kg q3w will be based on intrapatient dose escalation and DLT assessments as described below.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of consensus histologic, laboratory, and clinical diagnostic criteria of iMCD.
* Archival and/or baseline incisional/excisional biopsy for retrospective central histologic confirmation of iMCD.
* CDCNRC-defined disease progression on or after prior treatment with siltuximab at 11 mg/kg q3w without unacceptable toxicity within 12 weeks between the last dose of siltuximab and the date of signed patient informed consent form (ICF).
* At least 1 measurable abnormal lymph node mass that is ≥1 cm in its longest transverse diameter as assessed by computerized tomography (CT) scan that has not been previously irradiated.
* Elevated (>10 mg/L) and rising serum CRP in the absence of additional iMCD treatment.
* Evidence of at least an additional one of the following laboratory or clinical signs of iMCD per international, evidence-based consensus diagnostic criteria for HIV or HHV 8-negative iMCD:

  * Anemia, thrombocytopenia, hypoalbuminemia, renal dysfunction, or polyclonal hypergammaglobulinemia.
  * Constitutional symptoms (night sweats, fever (>38°C), weight loss, or fatigue (CTCAE lymphoma B-symptoms score ≥2), large spleen and/or liver, fluid accumulation, eruptive cherry hemangiomatosis/violaceous papules, or lymphocytic interstitial pneumonitis.
* Adequate clinical laboratory measurements within 3 weeks prior to study entry in all parameters below:

  * Absolute neutrophil count ≥1.0 × 109/L, hemoglobin <17 g/dL, and platelets ≥50 × 109/L without transfusion, hematopoietic growth factors, or both for >7 days prior to measurement.
  * AST, ALT, total bilirubin, and alkaline phosphatase ≤5 × ULN.
  * Fasting cholesterol <300 mg/dL and fasting triglyceride <400 mg/dL.
* Age ≥12 years.

Exclusion Criteria:

* Documentation of HIV or HHV-8 infection or presence of other infection-related disorders that resemble clinical or histological features of iMCD
* Diagnosis of any malignant/benign lymphoproliferative disorders
* Diagnosis of autoimmune/autoinflammatory disease
* Treatment with corticosteroids (prednisone dose-equivalent >1 mg/kg/day) within 7 days prior to study entry.
* History of solid organ transplant, allogeneic bone marrow transplant, or allogeneic peripheral blood stem cell transplant.
* Previous malignancy with the following exceptions:

  * Past malignancy with treatment that was completed at least 2 years before signing informed consent and the patient has no evidence of disease, or
  * Concurrent malignancy that is clinically stable and does not require tumor-directed treatment (eg, nonmelanoma skin cancer and carcinoma in situ)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Assess the Clinical Benefit Response (CBR) of Siltuximab | 12 Weeks
  Assess the clinical benefit response (CBR) of increased siltuximab doses in patients with IL-6-driven (C-reactive protein [CRP]-elevated and rising) idiopathic multicentric Castleman disease (iMCD) after disease progression on the standard siltuximab dose schedule. CBR defined as complete response (CR), partial response (PR), or stable disease (SD) lasting ≥12 weeks per Castleman Disease Collaborative Network Response Criteria (CDCNRC).

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of increased Siltuximab doses | 12 Weeks
  Incidence of Adverse Events (AEs), serious adverse events (SAEs), suspected unexpected serious adverse reactions (SUSARs), incidence of abnormal laboratory test results incidence of dose-limiting toxicities (DLTs)
Pharmacokinetics (Vd) | 12 Weeks
  To test the patient's drug propensity
Pharmacokinetics (CL) | 12 Weeks
  To test the volume of plasma cleared of drug per unit time
Pharmacokinetics (AUC) | 12 Weeks
  To test the extent of exposure to a drug and its clearance rate from the body
Pharmacokinetics (Cmin / Cmax) | 12 Weeks
  To test the minimum (Cmin) and the maximum (Cmax) blood plasma concentration
Pharmacokinetics (Ctrough) | 12 Weeks
  To test the minimum drug concentration after a dose
Pharmacokinetics (Tmax) | 12 Weeks
  To test the time taken to reach Cmax
Evaluate the efficacy of increased siltuximab doses after disease progression on prior siltuximab treatment. | 12 Weeks
  The primary efficacy endpoint is CBR defined as CR, PR, or SD lasting ≥12 weeks per CDCNRC based on evaluation of biochemical, lymph node, and symptom response
Evaluate the immunogenicity of increased siltuximab doses after disease progression on prior siltuximab treatment. | 12 Weeks
  Immunogenicity will be assessed through the detection of antibodies against siltuximab, and will be conducted via immunoassay ± serum IL-6 levels on Day 1 of Cycle 1, 3, 6 and every 4 cycles thereafter, before administration of siltuximab.
To evaluate the patient-reported outcomes (PROs) using the EQ-5D Instrument | 12 Weeks
  The secondary outcome measures will include the health status measures of the EuroQuality of Life Five Dimensions (EQ-5D) has the following dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the 5 dimensions
To evaluate the patient-reported outcomes (PROs) using the MCD-SS Instrument | 12 Weeks
  The Multicentric Castleman disease symptom score (MCD-SS) lists 10 symptoms which are graded on a scale: Did not experience (0); Very mild (2); Mild (4); Moderate (6); Severe (8); Very Severe (10). The mean score of the ten items is calculated and a higher score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Keuker, MD, Study Director — Syneos Health
Locations (1):
- Edward W. Sparrow Hospital, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No